CLINICAL TRIAL: NCT06508008
Title: Verification of the Effect of Intermittent Negative Pressure Sputum Suction Through Oral Pharyngeal Ventilation Tube in Comatose Patients
Brief Title: Rapid and Safe Sputum Suction Method Validation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Affiliated Hospital of Nantong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2024-K119-01
Record Dates: First submitted 2024-06-30; First posted 2024-07-18 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-06

CONDITIONS: Sputum

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intermittent negative pressure sputum suction through oral pharyngeal airway (Experimental): (1) Insert the oropharyngeal airway parallel into the oral cavity; (2) Apply paraffin oil to the front end of the sputum suction tube; (3) The suction tube is inserted into the deep oral cavity through the middle lumen of the oropharyngeal airway; (4) Intermittent negative pressure for suction and suction of sputum
  Interventions: Procedure: continuous negative pressure suction; Procedure: Intermittent negative pressure sputum suction through oral pharyngeal airway
- continuous negative pressure suction (No Intervention): (1) Use a tongue depressor to open the mouth; (2) Lubricating the front end of the sputum suction tube with paraffin oil; (3) Insert a suction tube into the oral cavity to aspirate phlegm.

INTERVENTIONS:
Procedure: continuous negative pressure suction — (1) Open the mouth with a tongue depressor; (2) Apply paraffin oil to the front end of the sputum suction tube; (3) Insert a suction tube into the mouth to aspirate phlegm.
  Arms: Intermittent negative pressure sputum suction through oral pharyngeal airway
Procedure: Intermittent negative pressure sputum suction through oral pharyngeal airway — (1) Insert the oropharyngeal airway parallel into the oral cavity; (2) Apply paraffin oil to the front end of the sputum suction tube; (3) The suction tube is inserted into the deep oral cavity through the middle lumen of the oropharyngeal airway; (4) Intermittent negative pressure for suction and suction of sputum
  Arms: Intermittent negative pressure sputum suction through oral pharyngeal airway

SUMMARY:
600 comatose patients admitted to the hospital in China from June 2024 to June 2028 were randomly divided into groups A and B. Group A used intermittent negative pressure suction through oral and pharyngeal ventilation, while group B used continuous negative pressure suction through regular oral and nasal suction.

DETAILED DESCRIPTION:
Research content: (1) Selection and placement methods of oropharyngeal ventilation tubes, studying the application effects of different models and sizes of oropharyngeal ventilation tubes in critically ill patients, exploring the best placement method to improve the efficiency and safety of sputum suction operations. (2) The norms and techniques of sputum suction, the steps, techniques, and precautions of sputum suction, the depth, strength, time of insertion, and when to interrupt negative pressure, in order to minimize damage to the patient's respiratory mucosa. (3) Evaluation of patient comfort and tolerance, assessing the tolerance and potential adverse reactions of critically ill patients during oral pharyngeal intubation for sputum suction, providing a basis for optimizing sputum suction. (4) Evaluation of sputum suction effect, comparing blood oxygen saturation, respiratory distress, sputum sounds, and other indicators before and after sputum suction to evaluate the effectiveness of sputum suction.

ELIGIBILITY:
Inclusion Criteria:

* 1. Clinical diagnosis of stroke; 2. Clinical diagnosis of comatose;

Exclusion Criteria:

* 1. Clinical diagnosis of multiple organ failure; 2. Clinical diagnosis of multiple organ bleeding;

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2024-02-18 (Actual); Primary Completion 2024-07-09 (Actual); Study Completion 2024-08-18 (Estimated)

PRIMARY OUTCOMES:
Blood oxygen saturation before and after sputum aspiration | Not exceeding 1 day
  The degree of binding between oxygen and hemoglobin (Hb) in arterial blood
Suctioning time | Not exceeding 2 minute
  All time required for sputum suction process
Degree of airway bleeding | Not exceeding 30 minute
  Use a disposable sputum collection device to aspirate sputum for patients and differentiate the blood content under a blue LED light.

SECONDARY OUTCOMES:
Patient family satisfaction | Not exceeding 1 day
  After suctioning, use a satisfaction questionnaire to survey the operating nurses, with a minimum score of 1 and a maximum score of 5. The higher the value, the higher the satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Tao Zhang, MD, Study Chair — Ethics Committee of Nantong University Affiliated Hospital
Locations (1):
- Affiliated Hospital of Nantong University, Nantong, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No